CLINICAL TRIAL: NCT07088900
Title: The Effectiveness of Dexmedetomidine as an Adjuvant for Bupivacaine Caudal Block in Pediatric Open Appendectomy Under General Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Tarek Hussein, doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MD352a/2023/2025
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: Appendectomy; Pediatric
Keywords: caudal; dexmedetomidine; open appendectomy
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients will receive a single-shot caudal block with 1 mL/kg of 0.25% bupivacaine mixed with 1 mL of normal saline.
  Interventions: Procedure: caudal block with bupivacaine
- Experimental Group (Experimental): Patients will receive a single-shot caudal block with 1 mL/kg of 0.25% bupivacaine mixed with 1 µg/kg of dexmedetomidine (diluted in 1 mL of normal saline).
  Interventions: Procedure: caudal block using dexmedetomidine with bupivacaine

INTERVENTIONS:
Procedure: caudal block using dexmedetomidine with bupivacaine — Patients will receive a single-shot caudal block with 1 mL/kg of 0.25% bupivacaine mixed with 1 µg/kg of dexmedetomidine (diluted in 1 mL of normal saline).
  Arms: Experimental Group
Procedure: caudal block with bupivacaine — Patients will receive a single-shot caudal block with 1 mL/kg of 0.25% bupivacaine mixed with 1 mL of normal saline
  Arms: Control Group

SUMMARY:
This study aims to evaluate if adding dexmedetomidine to bupivacaine in a caudal block can provide longer and better quality pain relief for children after open appendectomy surgery. The study will also assess the effect of this combination on the quality of recovery, including the incidence of emergence delirium, and its overall safety profile.

ELIGIBILITY:
inclusion criteria:

* ASA (American Society of Anesthesiologists) physical status I or II.
* Legal guardian provides written informed consent. Exclusion Criteria
* Refusal of participation by the legal guardian.
* Known allergy or hypersensitivity to local anesthetics or dexmedetomidine.
* Coagulation disorder or receiving anticoagulant therapy.
* Active infection at or near the injection site.
* Significant anatomical abnormalities of the lumbosacral spine.
* Pre-existing neurological disorders, psychiatric disorders, or a history of convulsions.
* Anticipated surgery time of more than 2.5 hours.
* Patients with severe asthma or active wheezing.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Time to First Rescue Analgesia: | Up to 24 hours post-caudal block
  Defined as the time interval in minutes from the performance of the caudal block until the first administration of rescue analgesia (ibuprofen), which is prompted by a FLACC pain score of ≥ 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university hospitals, Cairo, Egypt